CLINICAL TRIAL: NCT03237169
Title: Performance of a New REsting Pressure Index During Invasive Angiography Compared To Adenosine Hyperemic FFR
Acronym: PREDICT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centro Hospitalar Lisboa Ocidental (Other Government)
Collaborators: Abbott Medical Devices (Industry); Cardiovascular Research Foundation, New York (Other)
Responsible Party: Principal Investigator, Luis Raposo, Principal Investigator, Centro Hospitalar Lisboa Ocidental
Other Study IDs: 2017-02
Record Dates: First submitted 2017-07-31; First posted 2017-08-02 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Fractional Flow Reserve, Myocardial; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective cohort: Prospective cohort of patients with stable or stabilized coronary artery disease and de novo coronary lesions, in whom functional evaluation is performed, according do standard clinical indications.

SUMMARY:
To test the feasibility and diagnostic accuracy of a new automated pressure derived resting index (Pd/Pamin), using FFR as gold standard, in de novo coronary lesions in which invasive physiological evaluation is warranted.

DETAILED DESCRIPTION:
Coronary lesions with a potential indication for percutaneous coronary intervention or warranting invasive physiological interrogation (in the opinion of the investigator) will undergo PressureWire™ assessment under 2 conditions: rest and adenosine hyperemia. The measurements at rest (standard Pd/Pa and Pd/Pamin) will be repeated to assess test/retest repeatability. Subsequent treatment decisions will be made by the operator according to the standard practice based on the adenosine FFR value together with all other clinical information.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing FFR assessment for standard clinical indications, according to individual operator decision.
2. Age ≥ 18 years.
3. Provided signed written informed consent for data collection the collection.
4. De novo coronary artery disease in target vessel.
5. Single or multiple vessel disease.
6. Patient eligible for elective or ad hoc PCI (or CABG), if revascularization is deemed indicated, in the setting of stable coronary artery disease or non-culprit lesions of non-ST elevation acute coronary syndromes (only in deferred procedures).
7. Stenosis deemed amenable for both evaluation with a pressure wire and for potential revascularization.

Exclusion Criteria:

1. Subjects with restenosis in the target vessel.
2. Known severe renal insufficiency (examples being but not limited to eGFR <30 ml/kg/min, serum creatinine ≥ 2.5 mg/dL or on dialysis).
3. Aorto-ostial lesion location within 3 mm of the aorta junction (both right and left).
4. Vessel(s) and lesion(s) not amenable for evaluation with a PressureWire™ and/or revascularization.
5. Tandem lesions
6. Moderate lesions in patients with multivessel disease in whom at least one lesion in another major epicardic vessel is severe (to minimize lesion interaction), unless the severe lesion is treated first (see above).
7. Left ventricular ejection fraction <50%
8. Known severe left ventricular hypertrophy
9. Atrial fibrillation or any other significant arrhythmia (including an heart rate <50/min on sinus rhythm)
10. Systolic blood pressure <90 mmHg.
11. Any other medical condition that in the opinion of the investigator will interfere with patient safety or study results
12. Currently participating in another clinical study that interferes with study results.
13. Pregnant or nursing females
14. Planned or prior heart transplantation or listed for heart transplant.
15. Any condition that precludes the subject from undergoing PCI or any of the protocol mandated procedures, for example subjects with a prior history heparin induced thrombocytopenia, known intolerance to adenosine or with a contra-indication for dual anti-platelet therapy.
16. Patients with severe valvular disease
17. Patients with severe pulmonary disease
18. Culprit lesions in ACS patients are not to be included nor non-culprit lesions in patients with a recent STEMI undergoing staged procedures.
19. Patients with a CTO, regardless of the presence and the extent of angiographic collaterals from the target vessel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive subjects scheduled for coronary angiography or PCI in whom operator decides to perform FFR will be approached for enrollment. Being a first-in-man study of a novel pressure index intended for future validation and use in a clinical setting, a full assessment of its range throughout the entire spectrum of lesion severity is warranted. As such, the protocol will allow for the inclusion of both less severe as well as of critical (>90%) lesions. Patients with either single or multiple vessel disease will be included.
  Data on additional lesions may or may not be collected but will not be used in the study. Vessels with sequential stenosis and tandem lesions will be evaluated and treated according to routine clinical practice, but not included in the study data collected.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-10-28 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of Pd/Pamin vs FFR | baseline
  Agreement will be tested using the established FFR 0.8 threshold as the binary reference standard.

SECONDARY OUTCOMES:
Discriminative power of Pd/Pamin and the best cut-off, taking FFR as gold | baseline
  ROC analysis using FFR as reference
Feasibility of Pd/Pamin measurements | Baseline
  Description of how often can Pd/Pamin can be measured accurately

CONTACTS AND LOCATIONS:
Overall Officials: Luis Raposo, MD, Principal Investigator — Centro Hospitalar de Lisboa Ocidental; Sergio Bravo Baptista, MD, PhD, Study Chair — Hospital Fernando da Fonseca
Locations (6):
- St. Francis Hospital The Heart Center, New York, New York, United States
- Department of Cardiology, University Hospital, Lille, France
- Institute of Cardiology, Catholic University of the Sacred Heart, Rome, Italy
- Portugal (3):
  - Hospital Prof. Doutor Fernando da Fonseca, Amadora
  - Centro Hospitalar de Lisboa Ocidental - Hospital de Santa Cruz, Carnaxide
  - Centro Hospitalar de Lisboa Central (CHLC) - Hospital de Santa Marta, Lisbon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levine GN, Bates ER, Blankenship JC, Bailey SR, Bittl JA, Cercek B, Chambers CE, Ellis SG, Guyton RA, Hollenberg SM, Khot UN, Lange RA, Mauri L, Mehran R, Moussa ID, Mukherjee D, Nallamothu BK, Ting HH; American College of Cardiology Foundation; American Heart Association Task Force on Practice Guidelines; Society for Cardiovascular Angiography and Interventions. 2011 ACCF/AHA/SCAI Guideline for Percutaneous Coronary Intervention. A report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines and the Society for Cardiovascular Angiography and Interventions. J Am Coll Cardiol. 2011 Dec 6;58(24):e44-122. doi: 10.1016/j.jacc.2011.08.007. Epub 2011 Nov 7. No abstract available. PMID 22070834
- [Background] Task Force on Myocardial Revascularization of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS); European Association for Percutaneous Cardiovascular Interventions (EAPCI); Wijns W, Kolh P, Danchin N, Di Mario C, Falk V, Folliguet T, Garg S, Huber K, James S, Knuuti J, Lopez-Sendon J, Marco J, Menicanti L, Ostojic M, Piepoli MF, Pirlet C, Pomar JL, Reifart N, Ribichini FL, Schalij MJ, Sergeant P, Serruys PW, Silber S, Sousa Uva M, Taggart D. Guidelines on myocardial revascularization. Eur Heart J. 2010 Oct;31(20):2501-55. doi: 10.1093/eurheartj/ehq277. Epub 2010 Aug 29. No abstract available. PMID 20802248
- [Background] Mamas MA, Horner S, Welch E, Ashworth A, Millington S, Fraser D, Fath-Ordoubadi F, Neyses L, El-Omar M. Resting Pd/Pa measured with intracoronary pressure wire strongly predicts fractional flow reserve. J Invasive Cardiol. 2010 Jun;22(6):260-5. PMID 20516504
- [Background] Sen S, Escaned J, Malik IS, Mikhail GW, Foale RA, Mila R, Tarkin J, Petraco R, Broyd C, Jabbour R, Sethi A, Baker CS, Bellamy M, Al-Bustami M, Hackett D, Khan M, Lefroy D, Parker KH, Hughes AD, Francis DP, Di Mario C, Mayet J, Davies JE. Development and validation of a new adenosine-independent index of stenosis severity from coronary wave-intensity analysis: results of the ADVISE (ADenosine Vasodilator Independent Stenosis Evaluation) study. J Am Coll Cardiol. 2012 Apr 10;59(15):1392-402. doi: 10.1016/j.jacc.2011.11.003. Epub 2011 Dec 7. PMID 22154731
- [Background] Ganz P, Abben R, Friedman PL, Garnic JD, Barry WH, Levin DC. Usefulness of transstenotic coronary pressure gradient measurements during diagnostic catheterization. Am J Cardiol. 1985 Apr 1;55(8):910-4. doi: 10.1016/0002-9149(85)90716-7. PMID 3157307
- [Background] Gruntzig AR, Senning A, Siegenthaler WE. Nonoperative dilatation of coronary-artery stenosis: percutaneous transluminal coronary angioplasty. N Engl J Med. 1979 Jul 12;301(2):61-8. doi: 10.1056/NEJM197907123010201. PMID 449946
- [Background] Berry C, van 't Veer M, Witt N, Kala P, Bocek O, Pyxaras SA, McClure JD, Fearon WF, Barbato E, Tonino PA, De Bruyne B, Pijls NH, Oldroyd KG. VERIFY (VERification of Instantaneous Wave-Free Ratio and Fractional Flow Reserve for the Assessment of Coronary Artery Stenosis Severity in EverydaY Practice): a multicenter study in consecutive patients. J Am Coll Cardiol. 2013 Apr 2;61(13):1421-7. doi: 10.1016/j.jacc.2012.09.065. Epub 2013 Feb 6. PMID 23395076
- [Background] Ganz P, Harrington DP, Gaspar J, Barry WH. Phasic pressure gradients across coronary and renal artery stenoses in humans. Am Heart J. 1983 Dec;106(6):1399-406. doi: 10.1016/0002-8703(83)90052-2. PMID 6650363